CLINICAL TRIAL: NCT02417038
Title: Postoperative Respiratory Monitoring After Neuraxial Opioid Administration for Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Brendan Carvalho, Principle Investigator, Stanford University
Other Study IDs: 30189
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Depression
Keywords: Postoperative Respiratory Monitoring; Neuraxial Opioid Administration for Cesarean Delivery
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Capnostream — The Capnostream capnograph (is registered with the FDA) is supplied by Covidien. The Capnostream is a portable CO2 monitor with a pulse oximetry module to measure and record SpO2 (oxygen saturation) and heart rate continuously. The Capnostream provides waveform patterns for respiratory rate and EtCO2 measurement.
  Other Names: Capnograph

SUMMARY:
Respiratory depression occurs in labor and delivery; noticeably when neuraxial opioids are given.Pathophysiological respiratory depression -failure to respond to hypercapnia or hypoxia - is challenging to measure clinically.American Society of Anesthesiologist guidelines recommend suitable respiratory monitoring for 24 hours post cesarean delivery (CD).

Use of capnograph will enable us to assess breath-by-breathe respiration in a population receiving neuraxial opioids - potentially at risk for respiratory depression.

Our aim is to assess our ability to capture maternal postpartum respiratory parameters in a cohort following opioid neuraxial administration for CD.

DETAILED DESCRIPTION:
The investigators wish to test the efficacy of capnograph in detection of apnea and respiratory depression in women following cesarean delivery. Currently, routine intensive monitoring such as the investigators propose is not performed, and many apneas may go undetected.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status class I or II
* Age between 18 and 45
* Gestational age greater than 37 completed weeks
* Singleton pregnancy.

Exclusion Criteria:

* Contraindication for neuraxial analgesia (bleeding diathesis, neuropathy, severe scoliosis, previous spine surgery, local anesthetic allergy)
* Allergies to postoperative medication (opioids, NSAIDs, acetaminophen)
* Chronic opioid use
* Opioid administration in the previous 12 hours
* Inability to adequately understand the consent form
* Blocked nose or nasal deformity.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing cesarean delivery with neuraxial anesthesia.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2016-04-15 (Actual)

PRIMARY OUTCOMES:
CO2 monitoring | 24 hrs
  The Capnostream is a portable CO2 monitor with a pulse oximetry module to measure and record SpO2 and heart rate and provides waveform patterns for respratory rate and EtCO2 measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

REFERENCES:
- [Background] Clerici C. [Modifications of respiratory function during pregnancy]. Rev Pneumol Clin. 1999 Oct;55(5):307-11. French. PMID 10637899
- [Background] Kolarzyk E, Szot WM, Lyszczarz J. Lung function and breathing regulation parameters during pregnancy. Arch Gynecol Obstet. 2005 Jun;272(1):53-8. doi: 10.1007/s00404-004-0691-1. Epub 2004 Dec 23. PMID 15616844
- [Background] Trakada G, Tsapanos V, Spiropoulos K. Normal pregnancy and oxygenation during sleep. Eur J Obstet Gynecol Reprod Biol. 2003 Aug 15;109(2):128-32. doi: 10.1016/s0301-2115(03)00100-3. PMID 12860327
- [Background] Sultan P, Gutierrez MC, Carvalho B. Neuraxial morphine and respiratory depression: finding the right balance. Drugs. 2011 Oct 1;71(14):1807-19. doi: 10.2165/11596250-000000000-00000. PMID 21942973
- [Background] Grindheim G, Toska K, Estensen ME, Rosseland LA. Changes in pulmonary function during pregnancy: a longitudinal cohort study. BJOG. 2012 Jan;119(1):94-101. doi: 10.1111/j.1471-0528.2011.03158.x. Epub 2011 Oct 18. PMID 22004272
- [Background] Kato R, Shimamoto H, Terui K, Yokota K, Miyao H. Delayed respiratory depression associated with 0.15 mg intrathecal morphine for cesarean section: a review of 1915 cases. J Anesth. 2008;22(2):112-6. doi: 10.1007/s00540-007-0593-z. Epub 2008 May 25. PMID 18500606
- [Background] Pan PH, James CF. Anesthetic-postoperative morphine regimens for cesarean section and postoperative oxygen saturation monitored by a telemetric pulse oximetry network for 24 continuous hours. J Clin Anesth. 1994 Mar-Apr;6(2):124-8. doi: 10.1016/0952-8180(94)90009-4. PMID 8204230
- [Background] Wilson DL, Walker SP, Fung AM, O'Donoghue F, Barnes M, Howard M. Can we predict sleep-disordered breathing in pregnancy? The clinical utility of symptoms. J Sleep Res. 2013 Dec;22(6):670-8. doi: 10.1111/jsr.12063. Epub 2013 Jun 10. PMID 23745721
- [Background] Silva GE, Vana KD, Goodwin JL, Sherrill DL, Quan SF. Identification of patients with sleep disordered breathing: comparing the four-variable screening tool, STOP, STOP-Bang, and Epworth Sleepiness Scales. J Clin Sleep Med. 2011 Oct 15;7(5):467-72. doi: 10.5664/JCSM.1308. PMID 22003341
- [Background] Carvalho B. Respiratory depression after neuraxial opioids in the obstetric setting. Anesth Analg. 2008 Sep;107(3):956-61. doi: 10.1213/ane.0b013e318168b443. PMID 18713913
- [Derived] Weiniger CF, Akdagli S, Turvall E, Deutsch L, Carvalho B. Prospective Observational Investigation of Capnography and Pulse Oximetry Monitoring After Cesarean Delivery With Intrathecal Morphine. Anesth Analg. 2019 Mar;128(3):513-522. doi: 10.1213/ANE.0000000000003503. PMID 29958217